CLINICAL TRIAL: NCT00674037
Title: Efficacy of Monetary Incentives for Primary Care Physicians on Patients' Recruitment
Brief Title: Efficacy of Monetary Incentives for Primary Care Physicians on Patients
Acronym: COFRASAanc
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: default inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: P051042
Record Dates: First submitted 2008-04-09; First posted 2008-05-07 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2013-12

CONDITIONS: Recruitment
Keywords: recruitment; physicians participating in the recruitment of patients

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- inclusion with financial motivation (Experimental): 75 euros for each patient included
  Interventions: Other: monetary incentive
- no incentive (No Intervention): no incentive

INTERVENTIONS:
Other: monetary incentive — 75 euros for each patient included
  Arms: inclusion with financial motivation

SUMMARY:
Patients' recruitment is difficult in clinical trial. Financial incentives are frequently proposed to clinicians in private funded trials. However, the effect of these financial incentives has never been evaluated.

The purpose of this study is to evaluate the effect of financial incentive on the rate of recruitment of patients in a cohort study.

DETAILED DESCRIPTION:
Context: Patients' recruitment is difficult in clinical trials. Financial incentives are frequently proposed to clinicians in private funded trials. However, the effect of these financial incentives has never been evaluated.

Objective: to evaluate the effect of financial incentive on the rate of recruitment of patients in a cohort study.

Design: randomized controlled trial Setting: primary care Participants: physicians (GP and cardiologists) participating in the recruitment of patients in a cohort study (the COFRASA study). The COFRASA cohort study is including aortic stenosis aging patient.

Intervention:75 euros for each patient included Main outcome: percentage of physician including at least one patient at 3 months Secondary outcome: mean number of patients included at 6 months. Sample size 270 physicians

ELIGIBILITY:
Inclusion Criteria:

* Physicians participating in the COFRASA cohort study
* informed consent

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2006-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
number of patient included | 3 months

SECONDARY OUTCOMES:
number of patient included | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle BOUTRON, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Groupe hospitalier Bichat-Claude Bernard, Paris, France